CLINICAL TRIAL: NCT02507245
Title: Observational Longitudinal Study in Children Affected by Idiopathic Growth Hormone Deficiency (GHD): Lung Function Parameters Assessment; Quality of Life Assessment; Stress Parenting Assessment (Pneumo GHD)
Brief Title: Observational Longitudinal Study in Children Affected by Idiopathic Growth Hormone Deficiency (GHD)
Acronym: GHD
Status: Completed | Type: Observational
Sponsor: Stefania La Grutta, MD (Other)
Responsible Party: Sponsor-Investigator, Stefania La Grutta, MD, Stefania La Grutta, MD. Senior Researcher. Coordinator of Pediatric Allergy and Asthma Research Group. Institute of Biomedicine and Molecular Immunology, IBIM, National Research Council of Palermo, Italy., Istituto per la Ricerca e l'Innovazione Biomedica
Organization: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Other Study IDs: Verbale N°4/2013
Record Dates: First submitted 2015-06-03; First posted 2015-07-23 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Growth Hormone Deficiency
Keywords: GHD
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Growth Hormone-Releasing Hormone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- GHD Children: Treatment with Growth Hormone-Releasing Hormone in children affected by idiopathic growth hormone deficiency (GHD)
  Interventions: Drug: Growth Hormone-Releasing Hormone

INTERVENTIONS:
Drug: Growth Hormone-Releasing Hormone — From Baseline Visit (T0) to 6th Month Visit 0,025 mg/kg Growth Hormone/die. From 6th Month Visit to 12th Month Visit 0,030 mg/Kg Growth Hormone/die.
  Other Names: GH

SUMMARY:
The aim of this study is to assess the developmental patterns of lung function in children affected by growth hormone deficiency after one year of GH therapy.The assessment by specific questionnaires of quality of life and of parental stress index.Parameters will be evaluated at the time of the diagnosis and after 12 months of GH therapy.

DETAILED DESCRIPTION:
Observational longitudinal study in children affected by idiopathic growth hormone deficiency (GHD): lung function parameters assessment; quality of life assessment; stress parenting assessment (Pneumo GHD). The aim of this study is to assess the developmental patterns of lung function in children affected by growth hormone deficiency after one year of GH therapy.The assessment by specific questionnaires of quality of life and of parental stress index.Parameters will be evaluated at the time of the diagnosis and after 12 months of GH therapy.

ELIGIBILITY:
Inclusion Criteria:

* GH deficiency

Exclusion Criteria:

* Respiratory infections 4 weeks before the recruitment
* Children with autoimmune diseases
* Therapy with drugs able to modify the lung function

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 48 children affected by GH deficiency , recruited in the outpatient clinic of Pediatric Allergology & Pulmonology (PAP) of Respiratory Disease Research Center (RDRC) within the Institute of Biomedicine and Molecular Immunology (IBIM) of the National Research Council (CNR) of Palermo (RDRC-IBIM CNR), Italy.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2014-01; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Assessment of the developmental patterns of lung function before and after GH by spirometry | 1 year
  Assessment of lung function before and after administration of GH in children with growth hormone deficiency by spirometry